CLINICAL TRIAL: NCT01794065
Title: The Promus Element Rewards Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: REWARDS PE
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Stenosis
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Cypher: 100 patients who have received a Cypher stent during their coronary intervention
- Taxus Express: 100 patients who have received a Taxus Express stent during their coronary intervention
- Endeavor: 100 patients who have received an Endeavor stent during their coronary intervention
- Promus/Xience V: 100 patients who have received a Promus/Xience V stent during their coronary intervention
- Promus Element: 100 patients who have received a Taxus Element stent during their coronary intervention

SUMMARY:
This study is being done to study stent deformation on persons with de novo coronary lesions to determine how much deformation takes place and how often. The information gathered from the group that receives the Promus element stent will be compared to other groups that receive other contemporary drug eluting stents.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, 18 years or older;
* Patients with de-novo coronary lesions and slated to receive a Promus Element stent;
* Patients who are slated to undergo IVUS after stent deployment during implantation procedure

Exclusion Criteria:

* Patients receiving more than one drug-eluting stent within the same lesion during implantation procedure;
* Patients with in-stent restenosis;
* Patients who had IVUS imaging attained with manual pullback.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to receive a Promus Element stent implant, and have de novo coronary lesions.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Stent length | 1 day
  The primary endpoint of this study will be to assess the overall change in stent length post deployment by intravascualar ultrasound (IVUS) between the 5 stent groups.

SECONDARY OUTCOMES:
IVUS stent length | 1 day
  The secondary endpoints of this analysis will be to detect the occurrence of a 10% change in stent length by IVUS as compared to the labeled stent length.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Medstar Washington Hospital Center, Washington D.C., District of Columbia, United States